CLINICAL TRIAL: NCT05210465
Title: Objective Confirmation of thе Anti-ischemic Effectiveness of Trimetazidine 80mg Once Daily in Patients With Stable Angina Who Had a History of Myocardial Infarction (METHOD)
Acronym: METHOD
Status: Completed | Type: Observational
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-06795-067-RUS
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Dobutamine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with stable angina pectoris and prior MI
  Interventions: Other: speckle tracking mode of the stress ECHO test with dobutamine

INTERVENTIONS:
Other: speckle tracking mode of the stress ECHO test with dobutamine — speckle tracking mode of the stress ECHO test with dobutamine

SUMMARY:
METHOD is a prospective observational program that will be conducted in 1centre of the Russian Federation. Prospective follow-up will be for about 6 months. The METHOD study is a 2 visit study with first visit of inclusion and second visit of completion of the study. Patients with stable angina pectoris eligible to the study inclusion criteria will be invited to participate in this observational program. The parameters for analysis will be collected by doctors and entered into CRF. The final analysis will include data from patients who were taking TMZ 80 mg OD during the observational period. The decision to stop the study will be made once 36 patients receiving treatment with trimetazidine 80 mg OD will have been evaluated at V1.

It is expected that 5 cardiologists will participate in the program. The planned number of patients is 36.

DETAILED DESCRIPTION:
To describe antiischemic and antianginal effectiveness of trimetazidine OD 80 mg as well as adherence to the treatment with TMZ 80 mg OD in patients with stable angina pectoris and prior MI in real clinical practice in Russia

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 yearsAge older than 18 years
* Signed informed consent form
* Stable angina pectoris (CCS I-III FC) with signs of myocardial ischemia despite treatment with antianginal drug(s) present either clinically and/ or at stress ECHO test with dobutamine
* History of myocardial infraction occurred 6 months and more from the inclusion date
* Trimetazidine (TMZ) is recommended as add on to the current antianginal treatment and this recommendation precedes inclusion of a patient in the study
* Intention to perform a stress echo with spackle tracking precedes the start of TMZ
* Physician's intention to perform a stress ECHO test within a 6-month period after the date of inclusion in the study

Exclusion Criteria:

* Age over 75 years or under 18 years old
* Hypersensitivity to the active substance or any excipient specified in SmPc of TMZ 80 mg OD
* Parkinson's disease, parkinsonism symptoms, tremors, restless legs syndrome and other accompanying movement disorders
* Known severe or moderate renal impairment (creatinine clearance <60 ml / min).
* Angina pectoris of IV functional CCS class
* Heart failure IV functional class by NYHA
* Cardiac valves insufficiency with regurgitation of stage III and higher
* Myocardial infarction less than 6 months from the inclusion date
* Acute cerebrovascular event (stroke of various origins, transient ischemic attack) within 6 months before screening date
* Uncontrolled arterial hypertension of stage 3 (blood pressure above 180/100 mm Hg) despite ongoing antihypertensive therapy
* Fructose / sucrose intolerance, presence of glucose-galactose malabsorption syndrome, sucrose-somaltase deficiency and other enzymopathies associated with intolerance to sucrose, which is part of the drug
* Pregnancy, breastfeeding
* Any contraindications to stress echocardiography with dobutamine

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with stable angina pectoris and prior MI in real clinical practice in Russia
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
To describe antiischemic effectiveness of TMZ 80 mg OD assessed by the speckle tracking mode of the stress ECHO test with dobutamine in patients included in the study. | 6 months

SECONDARY OUTCOMES:
To describe antianginal effectiveness of TMZ 80 mg OD in patients included in the study | 6 months
To describe adherence to TMZ 80 mg OD in patients included in the study; | 6 months
To describe correlations between adherence (low, medium or high) to the treatment with TMZ 80 mg OD and antiischemic and antianginal effectiveness of TMZ 80 mg OD in patients included in the study; | 6 months
To describe impact on quality of life (QoL) to the treatment with TMZ 80 mg OD | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - "Institute for Complex Issues of Cardiovascular Diseases", Kemerovo
  - Barbarash Olga Leonidovna, Moscow